CLINICAL TRIAL: NCT05611021
Title: Acute Responses to Arm-Crank Exercise on Cardiovascular Function of Patients With Peripheral Artery Disease: Randomized Crossover Study
Brief Title: Acute Responses to Arm-Crank Exercise on Cardiovascular Function of Patients With Peripheral Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Marilia de Almeida Correia, PhD, University of Nove de Julho
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AcuteEBPAD
Record Dates: First submitted 2022-10-20; First posted 2022-11-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Intermittent Claudication; Cardiovascular Diseases; Blood Pressure; Endothelial Dysfunction; Peripheral Arterial Disease
MeSH Terms: conditions — Intermittent Claudication; Cardiovascular Diseases; Peripheral Arterial Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The patients will perform three experimental conditions, in randomized order (walking, arm-cranking and control). The exercise conditions will be composed of 15 bouts of 2 minutes exercise with an intensity equivalent to 13-15 on the Borg's subjective perceived exertion scale.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The outcomes assessor is blind for the condition performed by the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Walking Condition (Experimental): In the walking condition, the patients will perform fifteen bouts of two minutes of treadmill walking with an interval of two minutes between bouts, at an intensity equivalent to 13-15 on Borg's subjective perceived exertion scale. The condition will have a total of sixty minutes of duration.
  Interventions: Behavioral: Exercise
- Arm-Cranking Condition (Active Comparator): In the arm-cranking condition, the patients will perform fifteen bouts of two minutes of arm-cranking with an interval of two minutes between bouts, at an intensity equivalent to 13-15 on Borg's subjective perceived exertion scale. The condition will have a total of sixty minutes of duration.
  Interventions: Behavioral: Exercise
- Control Condition (Sham Comparator): The control condition will consist of resting in the standing position for thirty minutes. The patients will be instructed to rest in the sitting position for two minutes at periods equivalent to the intervals from the exercise conditions, totalling sixty minutes of duration.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Three conditions will be tested: Walking, arm-cranking and control condition.

SUMMARY:
The aim of this study is to analyze acute responses of arm-cranking exercise on cardiovascular function of peripheral arterial disease patients and compare it to the main exercise recommendation, walking exercise.

DETAILED DESCRIPTION:
Twenty patients with peripheral arterial disease and claudication symptoms will be recruited. The patients will perform three experimental conditions, in randomized order (walking, arm-cranking and control). The exercise conditions will be composed of 15 bouts of 2 minutes exercise with an intensity equivalent to 13-15 on Borg's Subjective Perceived Exertion Scale. During the experimental conditions (walking, arm-cranking and control) blood pressure, heart rate and cerebral blood velocity will be evaluated, along with perceived exertion and affective responses. Before and after experimental conditions, vascular function, blood pressure, heart rate variability, cerebral blood velocity, subjective perceived exertion and affective responses will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Peripheral arterial disease diagnosis;
* Age ≥ 40 years old;
* If a woman, be in menopause without the use of hormone replacement therapy;
* Do not be an active smoker;
* Be apt to perform exercise.

Exclusion Criteria:

* Any change in medication;
* Any health impairment that contraindicates the practice of physical exercise.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline in vascular function post-exercise in the brachial and femoral arteries. | Change from baseline at post-intervention, after 20 minutes.
  Vascular function will be measured in the supine position by the flow-mediated dilation (FMD) technique, through Doppler ultrasonography.

SECONDARY OUTCOMES:
Change from baseline in blood pressure post-exercise. | Change from baseline at post-intervention, after 10 minutes.
  Blood pressure will be measured by an automatic monitor.
Change from baseline in heart rate variability post-exercise. | Change from baseline at post-intervention, after 30 minutes.
  Autonomic modulation of the cardiovascular system will be measured by the heart rate variability (HRV) technique, by a heart rate monitor valid for this function.
Change from baseline in cerebral blood velocity post-exercise. | Change from baseline at 35 minutes after the beginning of the exercise.
  Cerebral blood velocity will be measured by a transcranial doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Marilia Correia, PhD, Principal Investigator — Nove de Julho University; Raphael Ritti-Dias, PhD, Study Chair — Nove de Julho University
Locations (1):
- Nove de Julho University, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data is planned to be made available after the completion of the study, if required.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Six months after the completion of the study.
Access Criteria: The data will be shared with certified researchers in the field.